CLINICAL TRIAL: NCT00980018
Title: An Exploratory Trial to Assess the Improvement of Chronic Low-grade Non-hematologic Adverse Events Experienced by Patients With Philadelphia Chromosome Positive (Ph+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP) Treated With Imatinib When Switched to Nilotinib Treatment
Brief Title: An Exploratory Trial to Assess the Improvement of Adverse Events in Chronic Myelogenous Leukemia Patients Treated With Imatinib When Switched to Nilotinib Treatment
Acronym: MACS0999
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107AUS17
Record Dates: First submitted 2009-09-16; First posted 2009-09-18 (Estimated); Results first posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: CML; Leukemia; Tasigna; nilotinib; AMN107; CML-CP; Chronic Phase
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nilotinib (Experimental): Participants received two 150 [a total of 300 mg at each dosing] mg nilotinib capsules twice daily (bid) orally every morning and every evening approximately 12 hours apart and two 200 mg capsules [a total of 400 mg at each dosing] for patients enrolled prior to Protocol Amendment 1).
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — Participants received two 150 [a total of 300 mg at each dosing] mg nilotinib capsules twice daily (bid) orally every morning and every evening approximately 12 hours apart and two 200 mg capsules [a total of 400 mg at each dosing] for patients enrolled prior to Protocol Amendment 1).
  Other Names: Tasigna, nilotinib, AMN107,

SUMMARY:
The purpose of this exploratory study will be to examine changes in chronic low grade chronic adverse events, measured by Common Terminology Criteria for Adverse Events (CTCAE) grading, when patients are switched from imatinib to nilotinib therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age
2. Eastern Cooperative Oncology Group (ECOG) 0, 1, or 2
3. Diagnosis of CML-CP associated with Bcr-Abl quantifiable by RQ-PCR (IS)
4. Patients must be an imatinib responder and achieved the following efficacy milestones as appropriate for the length of time on imatinib therapy as per protocol
5. CML-CP patients initiated on any dose of imatinib
6. Ability to provide written informed consent prior to any study related screening procedures being done

Exclusion Criteria:

1. Loss of CHR or cytogenetic response
2. Prior accelerated phase or blast phase CML
3. Previously documented T315I mutation
4. Presence of chromosomal abnormalities (trisomy 8) and/or clonal evolution other than Ph+.
5. Previous treatment with any other tyrosine kinase inhibitor except for imatinib.
6. Treatment with other investigational agents within 30 days of Day 1.
7. History of non-compliance to medical regimens or inability to grant consent.
8. Women who are pregnant, breast feeding, or of childbearing potential without a negative serum test at baseline. Male or female patients of childbearing potential unwilling to use contraceptive precautions throughout the trial and 3 months following discontinuation of study drug. Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential. Women of childbearing potential must have a negative serum pregnancy test prior to the first dose of nilotinib.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (22):
- United States (19):
  - Highlands Oncology Group, Fayetteville, Arkansas
  - Hematology Oncology Services of Arkansas SC, Little Rock, Arkansas
  - USC Norris Cancer Center LAC & USC Medical Center, Los Angeles, California
  - Southwest Cancer Care Murrieta, Poway, California
  - Rocky Mountain Cancer Centers RMCC - Aurora, Greenwood Village, Colorado
  - Florida Cancer Institute, New Port Richey, Florida
  - Cancer Centers of Florida PA Cancer Centers of FL-Orlando-4, Ocoee, Florida
  - Stroger Cook County Hospital John H. Stroger Hospital, Chicago, Illinois
  - St. Francis Hospital and Health Centers IndianaBlood&MarrowTransplantn, Beech Grove, Indiana
  - St. Agnes Hospital, Baltimore, Maryland
  - St. Louis University Cancer Center, St Louis, Missouri
  - Northwest Cancer Specialists Salmon Creek Office, Portland, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - The Jones Clinic, Germantown, Tennessee
  - Texas Oncology, P.A., Bedford, Texas
  - Presbyterian Hospital of Dallas TexasOncology@PresbyterianHosp, Dallas, Texas
  - Texas Oncology Texas Oncology - Sugar Land, Dallas, Texas
  - MD Anderson Cancer Center/University of Texas, Houston, Texas
  - Cancer Care Centers of South Texas / HOAST CCC of So. TX- San Antonio(2), San Antonio, Texas
- Canada (3):
  - Novartis Investigative Site, Brampton, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec

REFERENCES:
- [Derived] Cortes JE, Lipton JH, Miller CB, Busque L, Akard LP, Pinilla-Ibarz J, Keir C, Warsi G, Lin FP, Mauro MJ. Evaluating the Impact of a Switch to Nilotinib on Imatinib-Related Chronic Low-Grade Adverse Events in Patients With CML-CP: The ENRICH Study. Clin Lymphoma Myeloma Leuk. 2016 May;16(5):286-96. doi: 10.1016/j.clml.2016.02.002. Epub 2016 Feb 16. PMID 26993758
- See also: Related Info — http://NovartisClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 15 centers in US and 4 centers in Canada from 10-December-2009 (first patient first visit) to 27-December-2012 (last patient last visit).
Pre-assignment Details: A total of 68 patients were screened out of which 52 enrolled and 40 completed the full duration of treatment.
Period: Overall Study
Arm/Group | Nilotinib
Started | 52
Completed | 40
Not Completed | 12
Not completed — Adverse Event | 8
Not completed — Patient withdrew consent | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Safety Set : All participants who received at least one dose of study drug and had at least one post-baseline safety assessment.
Arm/Group | Nilotinib
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.7 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Improvement in Imatinib Related Chronic Low Grade Non Hematologic Adverse Event (AE) After Switch to Treatment With Nilotinib at End of Cycle 3
Description: A patient was considered improved if 50% or more of the chronic imatinib-related chronic low grade nonhematologic AEs showed improvement (a decrease in CTCAE [Common Terminology Criteria for Adverse Events] grade or complete resolution).
Time Frame: End of Cycles 1, 2, and 3
Population: Full Analysis Set (FAS): All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 52
Participants
  End of Cycle 1 | 37
  End of Cycle 2 | 43
  End of Cycle 3 | 44

2. Secondary Outcome: Percentage of Participants Achieving Complete Cytogenetic Response (CCyR) After Switching to Nilotinib for Participants Not Reporting CCyR at Baseline
Description: Time to complete cytogenetic response is defined as time from baseline to first time of CCyR as documented by bone marrow cytogenetics. Cytogenetic response was assessed as applicable by bone marrow cytogenetics 6, 12, and 18 months after starting imatinib therapy. Assess CCyR by bone marrow cytogenics
Time Frame: Cycles 1, 2, 6, 9, and 12
Population: FAS : All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 7
Participants
  Cycle 1 | 2
  Cycle 2 | 3
  Cycle 3 | 0
  Cycle 6 | 2
  Cycle 9 | 0
  Cycle 12 | 0

3. Secondary Outcome: Percentage of Participants Achieving Major Molecular Response (MMR) After the Switch in the Therapy for Participants Not Reporting MMR at Baseline
Description: Major Molecular Response (MMR) value at Molecular MD is designated a percentage, which is equivalent to a 3-log reduction from a standardized baseline value from the International Randomized Interferon versus STI571 (IRIS) study or 0.1% per International Scale (IS). Time to MMR is defined as time from baseline to first time of MMR as documented by RQ-PCR
Time Frame: Cycles 1,2,3,6,9,12
Population: FAS : All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 18
Participants
  Cycle 1 | 2
  Cycle 2 | 6
  Cycle 3 | 3
  Cycle 6 | 2
  Cycle 9 | 2
  Cycle 12 | 0

4. Secondary Outcome: Log Change in BCR-Abl Transcript Level From Baseline After the Switch Therapy
Description: Levels of BCR-ABL transcripts were determined by quantitative RQ-PCR testing of peripheral blood and analyzed at a central testing laboratory. Log reduction in BCR-ABL transcripts levels from the standardized baseline value will be calculated for each sample from the reported percent ratio of BCR-ABL transcripts versus control gene transcripts converted to a reference standard.
Time Frame: Cycles 1,2,3,6,9, and 12
Population: FAS: All participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: log change from Baseline
Arm/Group | Nilotinib
Number analyzed (Participants) | 52
log change from Baseline
  Cycle 1 | -0.177 (0.3665)
  Cycle 2 | -0.407 (0.5748)
  Cycle 3 | -0.540 (0.6960)
  Cycle 6 | -0.718 (0.9313)
  Cycle 9 | -0.844 (0.9130)
  Cycle 12 | -0.902 (0.9913)

5. Secondary Outcome: Duration of Complete Cytogenetic Response
Description: Duration of Complete Cytogenetic Response is defined as the time from first CCyR to first loss of CCyR as documented by bone marrow cytogenetics, or by FISH assay, whichever is earlier. The duration of CCyR begins on the day of enrollment for patients reporting CCyR at baseline.
Time Frame: 18 months of follow up from the first documented response
Population: FAS: All participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nilotinib
Number analyzed (Participants) | 52
days
  Participants with CCyR at baseline: number analyzed (Participants) | 45
  Participants with CCyR at baseline | 319.7 (143.03)
  Participants achieving CCyR on study: number analyzed (Participants) | 7
  Participants achieving CCyR on study | 266.3 (86.73)

6. Secondary Outcome: Time to Complete Cytogenetic Response in Participants Not Reporting at Baseline
Description: For time to CCyR, an event is defined as achievement of CCyR documented by bone marrow cytogenetics.
Time Frame: Cycle 12
Population: FAS: All participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nilotinib
Number analyzed (Participants) | 7
months | 1.9 [0.9 to 5.7]

7. Secondary Outcome: Duration of Major Molecular Response
Description: Duration of Major Molecular Response is defined as the time from first MMR to first loss of MMR as documented by RQ-PCR. The duration of MMR begins on the day of enrollment for patients reporting MMR at baseline.
Time Frame: 18 months of follow up from the first documented response
Population: FAS : All participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nilotinib
Number analyzed (Participants) | 49
days
  Participants with MMR at baseline: number analyzed (Participants) | 34
  Participants with MMR at baseline | 277.6 (166.88)
  Participants achieving MMR on study: number analyzed (Participants) | 15
  Participants achieving MMR on study | 208.3 (123.61)

8. Secondary Outcome: Time to Major Molecular Response (MMR) in Participants With MMR Absent at Baseline
Description: For time to MMR, an event is defined as achievement of MMR documented by RQ-PCR. Patients with MMR at the Screening RQ-PCR assay are counted as having time to MMR equal to 0.
Time Frame: Cycles 1,2,3,6,9,12
Population: FAS : All participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nilotinib
Number analyzed (Participants) | 18
months | 2.8 [1.8 to 5.8]

9. Secondary Outcome: Time to Optimal Imatinib-related Adverse Event Improvement
Description: Time to optimal improvement is defined as the time when the sum of the total CTCAE toxicity grades for a patient's chronic low-grade imatinib-related adverse events reaches its minimum value.
Time Frame: 18 months of follow up from the date of the first dose of study drug to the time to maximum decrease in CTCAE grade of these events
Population: FAS: All participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Nilotinib
Number analyzed (Participants) | 52
months | 1.9 [1.0 to 2.1]

ADVERSE EVENTS:
Time Frame: 18 months of follow up from the date of the first dose of study drug to the time to maximum decrease in CTCAE grade of these events
Description: The analysis was performed on safety set population defined as all participants who received study drug and had at least one post-baseline safety assessment.
Arm/Group | Nilotinib
All-Cause Mortality (participants affected / at risk) | 0/52
Serious Adverse Events (participants affected / at risk) | 9/52
Other Adverse Events (participants affected / at risk) | 49/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=52)
Cardiac arrest (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pancreatitis acute (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Vulval cellulitis (Infections and infestations) | 1
Wound infection bacterial (Infections and infestations) | 1
Wound infection staphylococcal (Infections and infestations) | 1
Cartilage injury (Injury, poisoning and procedural complications) | 1
Scapula fracture (Injury, poisoning and procedural complications) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Facial palsy (Nervous system disorders) | 1
Ovarian torsion (Reproductive system and breast disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Arteriosclerosis (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nilotinib (N=52)
Dry eye (Eye disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 8
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 6
Nausea (Gastrointestinal disorders) | 11
Chest pain (General disorders) | 3
Chills (General disorders) | 5
Fatigue (General disorders) | 17
Pyrexia (General disorders) | 3
Sinusitis (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 6
Lipase increased (Investigations) | 3
Weight decreased (Investigations) | 5
Anorexia (Metabolism and nutrition disorders) | 7
Decreased appetite (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 12
Bone pain (Musculoskeletal and connective tissue disorders) | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 4
Headache (Nervous system disorders) | 17
Hypoaesthesia (Nervous system disorders) | 3
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Alopecia (Skin and subcutaneous tissue disorders) | 7
Dry skin (Skin and subcutaneous tissue disorders) | 7
Night sweats (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 12
Rash (Skin and subcutaneous tissue disorders) | 17
Skin lesion (Skin and subcutaneous tissue disorders) | 4
Hot flush (Vascular disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No